CLINICAL TRIAL: NCT00325234
Title: A Randomized Phase II Study of Two Chemotherapy Regimens, Pemetrexed-Carboplatin, and Gemcitabine-Vinorelbine, in Anthracycline and Taxanes Pretreated Advanced Breast Cancer Patients
Brief Title: Pemetrexed-Carboplatin and Gemcitabine-Vinorelbine in Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10826; H3E-EW-S098 (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-05-10; First posted 2006-05-12 (Estimated); Results first posted 2011-05-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Pemetrexed; Carboplatin; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed/Carboplatin (Experimental): Pemetrexed 600 mg/m^2 was administered intravenously over approximately 10 minutes on Day 1.
  Carboplatin was given over approximately 30 minutes on Day 1 beginning after the end of the Pemetrexed infusion, consistent with a target of AUC (Area under the plasma drug concentration versus time curve) 5.0 mg*min/mL. The cycle of treatment was 21 days.
  Interventions: Drug: Pemetrexed; Drug: Carboplatin
- Gemcitabine/Vinorelbine (Active Comparator): Vinorelbine 30 mg/m^2 was given over approximately 6-10 minutes on Day 1 and Day 8. Gemcitabine 1200 mg/m^2 was given over approximately 30 minutes on Day 1 and Day 8 beginning after the end of the Vinorelbine infusion. The cycle of treatment was 21 days.
  Interventions: Drug: Gemcitabine; Drug: Vinorelbine

INTERVENTIONS:
Drug: Pemetrexed — 600 mg/m^2, administered intravenously (IV) every 21 days until disease progression or unacceptable toxicity.
  Other Names: LY231514; Alimta
  Arms: Pemetrexed/Carboplatin
Drug: Carboplatin — AUC 5 mg*min/mL, administered IV every 21 days until disease progression or unacceptable toxicity.
  Arms: Pemetrexed/Carboplatin
Drug: Gemcitabine — 1200 mg/m^2 gemcitabine, administered IV on day 1 and day 8 every 21 days until disease progression or unacceptable toxicity.
  Other Names: LY188011; Gemzar
  Arms: Gemcitabine/Vinorelbine
Drug: Vinorelbine — 30 mg/m^2 vinorelbine administered IV on day 1 and day 8 every 21 days until disease progression or unacceptable toxicity.
  Arms: Gemcitabine/Vinorelbine

SUMMARY:
The primary purpose of this study is to help answer the following research questions:

* whether the chemotherapy combination therapy Pemetrexed-Carboplatin or Gemcitabine-Vinorelbine can help participants with advanced breast cancer to make the tumor smaller or disappear and for how long
* to learn more about the side effects in each chemotherapy combination treatment arm
* to assess how participants with advanced breast cancer report health changes while receiving any of the chemotherapy combination arm

ELIGIBILITY:
Inclusion Criteria:

* Females with histologic or cytologic diagnosis of advanced breast cancer. Lesions should not be amenable to surgery or radiation of curative intent.
* Performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) performance status scale.
* One prior chemotherapy containing anthracyclines as (neo)adjuvant or palliative 1st-line treatment.
* One prior chemotherapy containing taxanes as (neo) adjuvant or palliative 1st-line treatment.
* Prior radiation therapy is allowed to less than 25% of the bone marrow. Participants must have recovered from the toxic effects of the treatment prior to study enrollment (except for alopecia). Prior radiotherapy must be completed 30 days before study entry. Lesions that have been radiated cannot be included as sites of measurable disease unless clear tumor progression has been documented in these lesions since the end of radiation therapy.
* At least one uni-dimensionally measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Positron emission tomography [PET] scans and ultrasounds may not be used.
* Antitumoral hormonal treatment must be discontinued prior to enrollment.
* Estimated life expectancy of at least 3 months.
* Participant compliance and geographic proximity that allow adequate follow-up.
* Adequate organ function
* Female participants of childbearing potential must test negative for pregnancy within 7 days of enrollment based on a urine and/or serum pregnancy test and agree to use a reliable method of birth control during and for 6 months following the last dose of study drug.
* Participants must sign an informed consent document.
* Female participants must be at least 18 years of age.

Exclusion Criteria:

* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Have previously completed or withdrawn from this study or any other study investigating Pemetrexed, Gemcitabine, Carboplatin or Vinorelbine
* Have received more than one line of chemotherapy in Metastatic Breast Cancer. Participants having received more than one combination of anthracycline plus taxane.
* Are pregnant or breast-feeding.
* Have serious concomitant systemic disorders (e.g., active infection) that, in the opinion of the investigator, would compromise the safety of the participant or compromise the participant's ability to complete the study.
* Have a prior malignancy other than breast cancer, carcinoma in situ of the cervix, or nonmelanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence.
* Are unable to interrupt aspirin or other nonsteroidal anti-inflammatory agents for a 5-day period (8-day period for long-acting agents such as piroxicam), unless the Creatinine Clearance is greater than or equal to 80 ml/min.
* Have central nervous system (CNS) metastases.
* Have clinically relevant (by physical exam) third-space fluid collections (for example, ascites or pleural effusions) that cannot be controlled by drainage or other procedures prior to study entry.
* Are unable or unwilling to take folic acid, vitamin B12 supplementation, or dexamethasone.
* Concurrent administration of any other antitumor therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2006-06; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon- Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- Germany (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gütersloh
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stuttgart
- Italy (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bergamo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Livorno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Meldola
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Giovanni Rotondo
- South Africa (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durban
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morningside
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pretoria
- Spain (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Girona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lleida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zaragoza
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Besevler/Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bornova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kayseri

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Pemetrexed/Carboplatin: Pemetrexed 600 mg/m^2 was administered intravenously over approximately 10 minutes on Day 1. Carboplatin was given over approximately 30 minutes on Day 1 beginning after the end of the Pemetrexed infusion, consistent with a target of AUC 5.0 mg*min/mL. The cycle of treatment was 21 days.
Period: Overall Study
Arm/Group | Pemetrexed/Carboplatin | Gemcitabine/Vinorelbine
Started | 69 | 66
Received At Least 1 Dose of Study Drug | 65 | 66
Completed | 0 | 0
Not Completed | 69 | 66
Not completed — Adverse Event | 10 | 7
Not completed — Death due to Study Disease | 1 | 0
Not completed — Entry Criteria Not Met | 1 | 2
Not completed — Subject Decision | 6 | 8
Not completed — Physician Decision | 17 | 12
Not completed — Progressive Disease | 34 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed/Carboplatin | Gemcitabine/Vinorelbine | Total
Number analyzed (Participants) | 69 | 66 | 135
Age Continuous [Mean (Standard Deviation); unit: years] | 51.9 (11.38) | 52.3 (10.40) | 52.1 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 66 | 135
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 67 | 61 | 128
  African | 1 | 3 | 4
  Hispanic | 0 | 1 | 1
  East Asian | 1 | 0 | 1
  West Asian | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Spain | 18 | 18 | 36
  Switzerland | 5 | 4 | 9
  Israel | 9 | 9 | 18
  Germany | 9 | 12 | 21
  Italy | 16 | 14 | 30
  Turkey | 5 | 3 | 8
  South Africa | 7 | 6 | 13
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — The Eastern Cooperative Oncology Group (ECOG) scales and criteria are used by doctors to assess disease progression, assess the patient's living ability, and determine prognosis. The scale is as follows:
  0-Fully active, able to carry on all pre-disease performance without restriction. 1-Restricted in activity but ambulatory and able to perform sedentary work. 2-Ambulatory but unable to work. Up and about > 50% of waking hours. 3-Capable of only limited selfcare, confined to bed or chair > 50% of waking hours. 4-Completely disabled. Cannot self care. Totally confined to bed or chair. 5-Dead
  participants
    ECOG 0 | 39 | 39 | 78
    ECOG 1 | 28 | 27 | 55
    ECOG 2 | 2 | 0 | 2
Hormonal Receptor Status [Number; unit: participants] — Hormone receptor status is a positive or negative measure of estrogen (ER) or progesterone (PR) hormone receptors found in cancer cells. In hormone receptor negative tumors, estrogen and/or progesterone are not present in cancer cells. In hormone receptor positive tumors, estrogen and/or progesterone hormone receptors are present in the cancer cells.
  participants
    Estrogen and Progesterone Negative | 19 | 21 | 40
    Estrogen and/or Progesterone Positive | 49 | 44 | 93
    Unknown | 1 | 1 | 2
Human Epidermal Growth Factor Receptor 2 (HER-2/Neu) [Number; unit: participants] — The Human Epidermal Growth Factor Receptor 2 plays an important role in cell growth and development. HER-2/Neu status is determined by an assay. A positive HER-2/Neu result indicates that HER-2 gene receptors are present; negative HER-2/Neu indicates the absence of HER-2 gene receptors.
  participants
    Positive | 12 | 13 | 25
    Negative | 53 | 49 | 102
    Not Performed | 0 | 1 | 1
    Unknown | 4 | 3 | 7
Tumor Differentiation Grade [Number; unit: participants] — Classification of tumors into one of four grades based upon how similar in appearance the tumor cells are to normal cells, and by how many tumor cells are dividing. The more tumor cells that are dividing, the greater likelihood of tumor growth and the higher the tumor grade. A lower tumor grade is associated with a better prognosis.
  Grade 1 - Well-Differentiated, Low cell division Grade 2 - Moderately Differentiated, Moderate cell division Grade 3 - Poorly Differentiated, High cell division Grade 4 - Undifferentiated, High cell division
  participants
    Grade I | 6 | 3 | 9
    Grade II | 25 | 27 | 52
    Grade III | 32 | 30 | 62
    Unknown | 6 | 6 | 12
Pathological Diagnosis [Number; unit: participants] — This measure is the specific diagnosis of breast cancer based upon pathological diagnosis.
  participants
    Carcinoma, Ductal, Breast | 64 | 54 | 118
    Carcinoma, Lobular, Breast | 4 | 5 | 9
    Carcinoma, Inflammatory, Breast | 1 | 3 | 4
    Carcinoma, Mixed Cell, Breast | 0 | 1 | 1
    Other | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate
Description: Participants with best overall response determined from complete response (CR) or partial response (PR) according to Response Criteria in Solid Tumors (RECIST) criteria. For CR or PR, best response must be confirmed. A second assessment performed at 28 days. Two determinations of CR before progression required for rate to=CR. Evaluations include: CR=Disappearance of lesions. PR=≥30% size decrease of lesions. Progressive Disease (PD)=≥20% size increase of lesions. Stable Disease (SD)=Not enough shrinkage for PR nor enough increase for PD. Overall Response Rate=PR+CR/Qualified Participants*100.
Time Frame: Baseline up to 30 days of follow-up after 21 cycles of treatment
Population: All randomized patients who qualified for tumor response analysis by the following criteria: Females with histologic or cytologic diagnosis of advanced breast cancer previously treated with anthracyclines and taxanes. No concurrent antitumor therapy. Presence of measurable disease as defined by RECIST. Treatment with at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pemetrexed/Carboplatin: Pemetrexed 600 mg/m^2 was administered intravenously over approximately 10 minutes on Day 1. Carboplatin was given over approximately 30 minutes on Day 1 beginning after the end of the Pemetrexed infusion, consistent with a target of AUC 5.0. The cycle of treatment was 21 days.
- Gemcitabine/Vinorelbine: Vinorelbine 30 mg/m^2 was given over approximately 6-10 minutes on Day 1 and Day 8. Gemcitabine 1200 mg/m^2 will be given over approximately 30 minutes on Day 1 and Day 8 beginning after the end of the Vinorelbine infusion. The cycle of treatment was 21 days.
Arm/Group | Pemetrexed/Carboplatin | Gemcitabine/Vinorelbine
Number analyzed (Participants) | 64 | 61
percentage of participants
  Overall Response | 26.6 [16.3 to 39.1] | 29.5 [18.5 to 42.6]
  Complete Response | 0.0 [0.0 to 5.6] | 3.3 [0.4 to 11.3]
  Partial Response | 26.6 [16.3 to 39.1] | 26.2 [15.8 to 39.1]
  Stable Disease | 35.9 [24.3 to 48.9] | 34.4 [22.7 to 47.7]
  Progressive Disease | 26.6 [16.3 to 39.1] | 27.9 [17.1 to 40.8]
  Unknown | 10.9 [4.5 to 21.2] | 8.2 [2.7 to 18.1]

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR-RECIST criteria of (Complete Response [CR =Disappearance of lesions] or Partial Response [PR=≥30% size decrease of lesions]) is defined as time from the date when measurement criteria are met for CR or PR until the date of first observation of progressive disease (PD) or death from study disease. For participants who die from causes other than study disease and without PD, DOR will be censored at the date of death. For participants who have not died as of the data cut-off date who are without PD, DOR was censored at last contact date.
Time Frame: Time of response to progressive disease (up to 19 months)
Population: All randomized participants with CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Carboplatin | Gemcitabine/Vinorelbine
Number analyzed (Participants) | 17 | 19
Months | 7.7 [4.2 to 12.2] | 7.5 [4.9 to 8.3]

3. Secondary Outcome: Time to Progressive Disease (PD)
Description: Time to PD is defined as the time from the date of study enrollment to the first documented date of PD or death from study disease. For participants who die from causes other than study disease and without PD, time to PD was censored at the date of death. For participants not known to have died as of the data cut-off date and do not have PD, time to PD was censored at the last contact date. For participants who received subsequent chemotherapy (after discontinuation from the study chemotherapy) prior to disease progression, time to PD was censored at the date of subsequent chemotherapy.
Time Frame: Baseline to measured PD (up to 25.1 months)
Population: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Carboplatin | Gemcitabine/Vinorelbine
Number analyzed (Participants) | 69 | 66
Months | 5.1 [4.1 to 8.0] | 5.6 [4.2 to 7.5]

4. Secondary Outcome: Time To Treatment Failure (TTTF)
Description: TTTF is defined as the time from date of study enrollment to the first documented date of death, PD, or study treatment discontinuation due to adverse event (AE). For participants not known to have discontinued as of the data cut-off date, TTTF is censored at the last contact date. For participants who discontinued for reasons other than death, PD, or AE, TTTF is censored at the date of discontinuation.
Time Frame: Baseline to end of treatment (up to 21.9 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Carboplatin | Gemcitabine/Vinorelbine
Number analyzed (Participants) | 69 | 66
Months | 4.8 [3.3 to 7.0] | 5.1 [3.5 to 6.3]

5. Secondary Outcome: Time to Response
Description: Time to response (Complete Response(CR) or Partial Response (PR) is defined as the time from the date of study enrollment to the first date when the measurement criteria are met for complete response or partial response (whichever status is recorded first). CR=Disappearance of target lesions lesions. PR=≥30% size decrease of lesions.
Time Frame: Baseline to response (up to 7.8 months)
Population: All randomized participants with CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pemetrexed/Carboplatin | Gemcitabine/Vinorelbine
Number analyzed (Participants) | 17 | 19
Months | 1.8 [1.6 to 3.3] | 1.8 [1.6 to 3.1]

6. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: A listing of adverse events is presented in the Reported Adverse Event Module.
Time Frame: every cycle up to twenty-one 21-day cycles (plus 30 days of follow-up)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Pemetrexed/Carboplatin | Gemcitabine/Vinorelbine
Number analyzed (Participants) | 65 | 66
participants
  Adverse Events | 64 | 66
  Serious Adverse Events | 18 | 22

ADVERSE EVENTS:
Arm/Group | Pemetrexed/Carboplatin | Gemcitabine/Vinorelbine
Serious Adverse Events (participants affected / at risk) | 18/65 | 22/66
Other Adverse Events (participants affected / at risk) | 64/65 | 66/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Carboplatin (N=65) | Gemcitabine/Vinorelbine (N=66)
Anaemia (Blood and lymphatic system disorders) | 5 (10) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (6) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (10) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Medical device complication (General disorders) | 0 (0) | 1 (1)
Performance status decreased (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed/Carboplatin (N=65) | Gemcitabine/Vinorelbine (N=66)
Anaemia (Blood and lymphatic system disorders) | 32 (46) | 28 (36)
Leukopenia (Blood and lymphatic system disorders) | 28 (79) | 35 (84)
Lymphopenia (Blood and lymphatic system disorders) | 10 (13) | 8 (15)
Neutropenia (Blood and lymphatic system disorders) | 37 (120) | 51 (154)
Thrombocytopenia (Blood and lymphatic system disorders) | 17 (34) | 11 (23)
Palpitations (Cardiac disorders) | 1 (1) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 9 (12)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 10 (13)
Constipation (Gastrointestinal disorders) | 18 (24) | 26 (41)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 12 (14)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 4 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 31 (48) | 23 (73)
Stomatitis (Gastrointestinal disorders) | 7 (8) | 11 (12)
Vomiting (Gastrointestinal disorders) | 15 (20) | 15 (19)
Asthenia (General disorders) | 14 (23) | 13 (19)
Fatigue (General disorders) | 23 (38) | 26 (39)
Oedema peripheral (General disorders) | 6 (6) | 6 (7)
Pyrexia (General disorders) | 5 (6) | 21 (33)
Alanine aminotransferase increased (Investigations) | 11 (16) | 21 (30)
Aspartate aminotransferase increased (Investigations) | 9 (14) | 17 (25)
Blood alkaline phosphatase increased (Investigations) | 7 (7) | 7 (8)
Gamma-glutamyltransferase increased (Investigations) | 4 (4) | 11 (16)
Weight decreased (Investigations) | 3 (3) | 8 (8)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 12 (13)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (6) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (17)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6)
Dizziness (Nervous system disorders) | 5 (7) | 4 (4)
Dysgeusia (Nervous system disorders) | 3 (3) | 4 (4)
Headache (Nervous system disorders) | 7 (10) | 11 (16)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3) | 9 (14)
Anxiety (Psychiatric disorders) | 1 (1) | 6 (6)
Insomnia (Psychiatric disorders) | 6 (6) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 16 (16)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (11) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 9 (10)
Phlebitis (Vascular disorders) | 0 (0) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days